CLINICAL TRIAL: NCT00444730
Title: Urology Database for Outcomes Research
Status: Completed | Type: Observational
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2007-031
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer; Pelvic Pain; Incontinence
Keywords: Prostate Cancer; Prostatectomy; Pelvic pain; urgency; incontinence; frequency
MeSH Terms: conditions — Prostatic Neoplasms; Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Radical Prostatectomy — Surgical procedure for prostate cancer.
Procedure: InterStim Implantation — surgical placement of the interstim
  Other Names: interstim
Procedure: Pelvic organ prolapse repair — Surgical pelvic organ prolapse repair
  Other Names: prolapse repair

SUMMARY:
The purpose of initiating the urology database is to collect relevant retrospective data via chart review related to patients undergoing radical prostatectomy via the retropubic, perineal, laparoscopic, and robotic assisted laparoscopic approaches and InterStim implantation. This data will be utilized to evaluate the health benefits and outcomes of each of these procedures to enhance care and treatment.

DETAILED DESCRIPTION:
The objective of this study is to initiate and maintain a patient information database that will be used to study the impact of each surgical procedure on patients' overall health, quality of life, and bowel/bladder/sexual function.

The study coordinator will, on an ongoing basis, abstract needed medical information from inpatient hospital and physician office records for inclusion into the database.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing radical prostatectomy or InterStim implantation at William Beaumont Hospital.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing radical prostatectomy or InterStim implantation at William Beaumont Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2007-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States